CLINICAL TRIAL: NCT07180225
Title: Manual Therapy Combined With Breathing Exercises in Management of Rotator Cuff Impingement Syndrome
Brief Title: Manual Therapy Combined With Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Assoc. Prof, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-240-5
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Injuries
Keywords: breathing exercises; manual therapy; conventional therapy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: PARTICIPANTS ARE MASKED
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP I (Experimental): Participants received conventional TENS applied to painful points in the shoulder region. Following TENS, patients performed a physiotherapist-supervised exercise program.At the beginning of the treatment, participants were provided with normal range of motion exercises and isometric strengthening exercises.Also, Glenohumeral joint (GH) distraction, glenohumeral joint inferior gliding, anterior gliding, and posterior gliding, scapulothoracic joint distraction, scapulothoracic joint superior, inferior, medial, and lateral gliding techniques were added.
  Interventions: Other: Conventional therapy+manual therapy
- GROUP II (Experimental): In addition to the treatment program applied in Group 1, participants in the intervention group received the following: Glenohumeral joint (GH) distraction, glenohumeral joint inferior gliding, anterior gliding, and posterior gliding, scapulothoracic joint distraction, scapulothoracic joint superior, inferior, medial, and lateral gliding, diaphragmatic breathing exercises, pursed-lip breathing exercises, and relaxation breathing exercises.
  Interventions: Other: Conventional therapy+manual therapy+breathing exercises

INTERVENTIONS:
Other: Conventional therapy+manual therapy — Conventional therapy contains TENS and physiotherapist-supervised exercise program. These exercises are Wand exercises (15 repetitions each), codman exercises (1 minute in each direction), shoulder wheel exercises (5 minutes total), finger ladder exercises (10 repetitions), isometric exercises (10 repetitions each), capsular stretching exercises (10 repetitions each), pectoral muscle stretching and stabilization exercises (10 repetitions), shoulder stabilization exercises (5 minutes total), and strengthening exercises for the shoulder flexor, extensor, abductor, adductor, internal rotator, and external rotator muscles (15 repetitions each). In addition to them, manual therapy were applied to the shoulder region.
  Arms: GROUP I
Other: Conventional therapy+manual therapy+breathing exercises — In addition to the treatment program of Group I, breathing exercises were added. Each manual therapy technique was performed with 10 repetitions per participant. Similarly, participants were instructed to perform each breathing exercise with 10 repetitions. They were also asked to continue the breathing exercises at home, performing them three times a day with 10 repetitions per session for a duration of six weeks.
  Arms: GROUP II

SUMMARY:
Rotator cuff impingement syndrome is one of the most common causes of shoulder pain and functional limitation, with manual therapy frequently employed in its management. This study aimed to investigate the additional effects of incorporating breathing exercises into manual therapy on pain and function.

DETAILED DESCRIPTION:
Rotator cuff impingement syndrome is one of the most common causes of shoulder pain and functional limitation, with manual therapy frequently employed in its management. This study aimed to investigate the additional effects of incorporating breathing exercises into manual therapy on pain and function. The study was conducted with fifty-two individuals aged 18-65 diagnosed with rotator cuff impingement syndrome. Individuals who met the inclusion criteria were randomly and equally assigned to two groups. Participants in the control group received the cold pack, TENS, and conventional exercise program. Participants in the intervention group received manual therapy combined with respiratory exercises in addition to this therapy program. All participants received therapy three times a week for a total of six weeks. The Visual Analog Scale (VAS) and Shoulder Pain and Disability Index (SPADI), shoulder range of motion (ROM) assessments, and a spirometer were used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* being between 18 and 65 years of age;
* the presence of at least one of the following clinical findings: positive Neer Impingement Test, positive Hawkins-Kennedy Impingement test, or painful arc during active abduction or flexion
* experiencing pain in at least one of the resisted tests for internal rotation, external rotation, abduction, or flexion
* being able to participate in the face-to-face treatment program consisting of a total of 18 sessions

Exclusion Criteria:

* a history of upper extremity fracture; undergoing shoulder surgery on the affected side within the past 12 months
* significant shoulder weakness or loss of active shoulder function; the presence of systemic musculoskeletal disorders
* symptom reproduction during active or passive cervical movements; the presence of consciousness disorders, cognitive impairments; and having any diagnosed cardiovascular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | Baseline and 6 weeks
  Pain intensity was assesed with visual anaolg scale (VAS) that is a tool commonly used to assess the intensity of musculoskeletal pain. The VAS was used to evaluate the level of shoulder pain experienced by participants at rest, and during activity. Participants were asked to rate their pain intensity on a scale ranging from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst possible pain." The participants' responses were recorded in the case report forms
Disability | Baseline and 6 weeks
  Shoulder Pain and Disability Index (SPADI) is a self-reported, shoulder specific questionnaire developed to assess pain intensity and disability levels in individuals with musculoskeletal shoulder pain.The disability subscale includes eight items, where patients rate the difficulty, they experienced while performing daily activities in the past week, using a scale from 0 (no difficulty) to 10 (so difficult that assistance is required). The total SPADI score was calculated by converting the total raw score into a percentage. The final score ranges from 0 to 100, with higher scores indicating greater levels of pain and disability
Range of motion evaluation | Baseline and 6 weeks
  A universal goniometer was used to measure the shoulder joint's ROM in flexion, extension, abduction, internal rotation, and external rotation. Measurements were recorded in degrees. Each movement was performed three times, and the average of these three measurements was used for analysis. After each measurement, the participant returned their arm to the neutral position before the next repetition. The normal ROM values for the shoulder joint are as follows: 0-180° for flexion and abduction, 0-45° for extension and adduction, and 0-90° for internal and external rotation
Pulmonary system evaluation | Baseline and 6 weeks
  A firstMed SP-10 electronic handheld spirometer was used to evaluate respiratory function. Each participant was instructed to place a disposable mouthpiece between their lips and teeth, ensuring no air escaped. They were then encouraged to perform a rapid and deep inspiration followed immediately by a forceful and complete expiration. Participants were expected to exhale for at least 6 seconds. The test was terminated once adequate expiration was achieved. Among at least three properly performed consecutive trials, the highest value was recorded

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, PhD, Principal Investigator — İstanbul Medipol university; ŞULE AYAN, Principal Investigator — İstanbul Medipol university
Locations (1):
- Merve Yilmaz Menek, Istanbul, Turkey (Türkiye)